CLINICAL TRIAL: NCT00726661
Title: An Observational Study of Treatment Patterns and Safety Outcomes for Metastatic or Locally Recurrent Breast Cancer
Brief Title: An Observational Study of Treatment Patterns and Safety Outcomes for Metastatic or Locally Recurrent Breast Cancer (VIRGO)
Acronym: VIRGO
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AVF4349n
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; Locally Recurrent Breast Cancer; Avastin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and tissue

GROUPS / COHORTS (2):
- Chemotherapy Cohort: Eligible participants with HER2-negative disease who received their first cytotoxic chemotherapy and/or targeted therapy were observed until death, withdrawal of consent, loss to follow-up, or until study closure, whichever was sooner (approximately 4.5 years).
- Hormonal Therapy Cohort: Eligible participants with hormone receptor positive disease who received their first hormonal therapy for advanced disease were observed until death, withdrawal of consent, loss to follow-up, or until study closure, whichever was sooner (approximately 4.5 years).

SUMMARY:
This is a multicenter, prospective observational cohort study (OCS) designed to follow patients with locally recurrent or metastatic breast cancer in the United States. Two cohorts will be included:

* Patients with human epidermal growth factor receptor 2-negative (HER2-negative) disease receiving their first cytotoxic chemotherapy and/or targeted therapy (approximately 825 patients)
* Patients with hormone receptor-positive (HR-positive) disease receiving their first hormonal therapy for advanced disease (approximately 425 patients)

Patients who have received any chemotherapy for advanced disease more than 8 weeks prior to enrollment to this OCS will not be eligible. A total of approximately 1,250 patients will be enrolled. Approximately 150 study sites will be activated in order to achieve complete enrollment by December 2010.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Locally recurrent or metastatic breast cancer
* Receipt of first systemic cytotoxic chemotherapy and/or targeted therapy among those with HER2-negative disease or first hormone therapy among those with HR-positive disease for the treatment of locally recurrent or metastatic disease, within 8 weeks prior to enrollment

Exclusion Criteria

* Any medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to provide informed consent or comply with the treatment
* Any prior chemotherapy started more than 8 weeks prior to enrollment for the treatment of locally recurrent or for metastatic breast cancer
* Concurrent participation only in a blinded clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer clinic
Sampling Method: Non-Probability Sample
Enrollment: 1287 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 01 June 2008 to 31 December 2012 in the United States. A total of 1287 participants were enrolled.
Pre-assignment Details: Out of 1287 participants, 20 were not eligible for the study and were excluded. Of 1267 participants, 832 were observed in Chemotherapy cohort and 435 were observed in Hormonal Therapy cohort.
Groups:
- Chemotherapy Cohort: Eligible participants with human epidermal growth factor receptor 2-negative (HER2-negative) disease who received their first cytotoxic chemotherapy and/or targeted therapy were observed until death, withdrawal of consent, loss to follow-up, or until study closure, whichever was sooner (approximately 4.5 years).
Period: Overall Study
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort
Started | 832 | 435
Completed | 18 | 17
Not Completed | 814 | 418
Not completed — Lost to Follow-up | 36 | 11
Not completed — Withdrawal by Subject | 17 | 13
Not completed — Trial terminated by sponsor | 214 | 187
Not completed — Death | 475 | 159
Not completed — Physician Decision | 25 | 13
Not completed — Other | 47 | 35

BASELINE CHARACTERISTICS:
Population: Baseline characteristics was analyzed for all enrolled participants in respective individual groups (CT Cohort and HT Cohort); therefore, the data for 'mean age' for total population is not applicable for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort | Total
Number analyzed (Participants) | 832 | 435 | 1267
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.40 (11.98) | 63.99 (12.57) | 59.66 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 826 | 434 | 1260
  Male | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from enrollment to progression or death of any cause, whichever came first. The disease response status was assessed by the investigator according to the method of his or her choice. The choices included computed tomography (CT) scan, magnetic resonance imaging (MRI), bone scan, X-ray, Positron emission tomography (PET) or CT PET, physical exam, laboratory exam, and other method.
Time Frame: Approximately 4.5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort
Number analyzed (Participants) | 832 | 435
months | 8.54 [8.02 to 9.20] | 12.88 [10.81 to 14.69]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from enrolment to death of any cause.
Time Frame: Approximately 4.5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort
Number analyzed (Participants) | 832 | 435
months | 23.92 [22.24 to 26.71] | 44.78 [39.85 to NA] — Upper limit of confidence interval was non-estimable because of immaturity of follow-up.

3. Secondary Outcome: Number of Participants With Tumor Response
Description: The tumor response was measured as complete response, partial response, stable disease, progressive disease, or clinical deterioration based on their best overall response. The tumor response was assessed by the investigator according to the method of his or her choice. The choices included computed tomography (CT) scan, magnetic resonance imaging (MRI), bone scan, X-ray, Positron emission tomography (PET) or CT PET, physical exam, laboratory exam, and other method.
Time Frame: Approximately 4.5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort
Number analyzed (Participants) | 832 | 435
participants
  Complete response | 133 | 34
  Partial response | 259 | 107
  Stable disease | 226 | 180
  Progressive disease | 148 | 86
  Clinical deterioration | 2 | 0

4. Secondary Outcome: Number of Hormone Receptor-positive Participants Who Initiated Cytotoxic Chemotherapy Following Discontinuation
Description: Participants were assessed quarterly for progressive events and treatment status.
Time Frame: Approximately 4.5 years
Population: All enrolled participants in Hormonal Therapy Cohort were considered for this outcome measure. n = number of participants evaluated at that particular time point.
Measure: Number; unit: participants
Arm/Group | Hormonal Therapy Cohort
Number analyzed (Participants) | 435
participants
  First quarter (n = 93) | 37
  Second quarter (n = 91) | 40
  Third quarter (n = 81) | 39
  Fourth quarter (n = 92) | 45
  Fifth quarter (n = 99) | 45
  Sixth quarter (n = 83) | 44

5. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Events, Any AEs Leading to Early Treatment Discontinuation, and Adverse Events Leading to Hospitalization or Death
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An Serious Adverse Events (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Approximately 4.5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort
Number analyzed (Participants) | 832 | 435
participants
  Any AEs | 46 | 13
  Any SAEs | 76 | 22
  Any AEs leading to early treatment discontinuation | 89 | 19
  AEs leading to hospitalization or death | 67 | 20

6. Secondary Outcome: Number of Participants With Arterial Thromboembolic Events, Venous Thromboembolic Events, Left Ventricular Systolic Dysfunction, and Peripheral Neuropathy
Description: All AEs were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3 as Grade 1 (mild), Graded 2 (moderate), Grade 3 (severe), Grade 4 (very severe, life threatening, or disabling), and Grade 5 (death related to AE). Venous Thromboembolic Events (VTEs) included all Grade 4 or of more severity of deep vein thrombosis, pulmonary embolus; Arterial Thromboembolic Events (ATEs) Included new or worsening angina pectoris, myocardial infarction, stroke, transient ischemic attack, peripheral arterial ischemia of any NCI CTCAE grade; Left Ventricular Systolic Dysfunction (LVSD) included congestive heart failure) of NCI CTCAE Grade 2 or of more severity; Peripheral Neuropathy (PN) included sensory and/or motor events of Grade 3 or of more severity.
Time Frame: Approximately 4.5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort
Number analyzed (Participants) | 832 | 435
participants
  ATE (any Grade) | 10 | 5
  VTE (Grade >= 4) | 14 | 6
  LVSD (Grade >= 2) | 16 | 4
  PN (Grade >= 3) | 17 | 3

ADVERSE EVENTS:
Time Frame: Approximately 4.5 years
Description: SAEs and other AEs were collected for all enrolled participants.
Arm/Group | Chemotherapy Cohort | Hormonal Therapy Cohort
Serious Adverse Events (participants affected / at risk) | 76/832 | 22/435
Other Adverse Events (participants affected / at risk) | 46/832 | 13/435
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy Cohort (N=832) | Hormonal Therapy Cohort (N=435)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Bilateral subdural hematoma (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenic fever (Blood and lymphatic system disorders) | 1 | 0
Neutropenic sepsis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Acute systolic heart failure (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary arrest (Cardiac disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 4 | 0
Coronary artery ischemia (Cardiac disorders) | 1 | 0
Heart attack (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0
Left ventricular systolic dysfunction (Grade >=2) (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Grade 3) (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Grade 4) (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Pericardial effusion with impending tamponade (Cardiac disorders) | 0 | 1
Recurrent transient ischemic attack (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Intractable nausea (Gastrointestinal disorders) | 1 | 0
Perforated diverticulum (Gastrointestinal disorders) | 1 | 0
Perforation colon (Grade 1) (Gastrointestinal disorders) | 1 | 0
Persistant vomiting (Gastrointestinal disorders) | 1 | 0
Rectal bleeding (Gastrointestinal disorders) | 1 | 0
Viral gastroenteritis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Hospitalization for weakness that ended in death (cause unknown) (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Weakness (General disorders) | 1 | 0
Hepatic insufficiency related to metastatic breast cancer (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Infection peritioneal cavity (Infections and infestations) | 1 | 0
Infection-left breast (Infections and infestations) | 1 | 0
Line associated bacteremia (vascular chest port infection) (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 0 | 1
Severe thrush (Infections and infestations) | 1 | 0
Femoral neck fracture right hip (Injury, poisoning and procedural complications) | 1 | 0
Intertrochanteric hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Febrile neutropenia (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypercalcemeia (Metabolism and nutrition disorders) | 1 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain musculoskeletal joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathologic fracture of the femur (Musculoskeletal and connective tissue disorders) | 0 | 1
T4 intramedullary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute left occipital infarct (Nervous system disorders) | 0 | 1
Cord compression (Nervous system disorders) | 1 | 0
Hemorrhagic mass in brain (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 0
Peripheral neuropathy (Nervous system disorders) | 1 | 0
Posterior reversible encephtalopathy syndrome (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Acute renal failure (Renal and urinary disorders) | 1 | 0
Polyneuropathy (Renal and urinary disorders) | 1 | 0
Acute pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bilateral pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (nose hemorrhage) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Left lung atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolization (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bilateral leg ulcers (Skin and subcutaneous tissue disorders) | 1 | 0
Cellulitis of the left upper extremity (Skin and subcutaneous tissue disorders) | 1 | 0
Left heel ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thromboembolic events (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Elevated blood pressure (Vascular disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Moderate size infarct involving a portion of the right middle cerebral artery territory (Vascular disorders) | 1 | 0
Multi-organ failure (shock) (Vascular disorders) | 0 | 1
Severe venous thromboembolic event (Grade > =4) (Vascular disorders) | 1 | 0
Stroke (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Thrombosis/embolism (Vascular disorders) | 1 | 0
Thrombosis/thrombus/embolism - pulmonary embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy Cohort (N=832) | Hormonal Therapy Cohort (N=435)
Left ventricular systolic dysfunction (Grade >=2) (Cardiac disorders) | 5 | 3
Congestive heart failure (Cardiac disorders) | 1 | 0
Decreased ejection fraction (Cardiac disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Worsening anemia (Blood and lymphatic system disorders) | 1 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Intermittent nosebleeds grade 1 (Investigations) | 1 | 0
Malignant pleural effusion indicating disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0
Arterial thromboembolic event (Vascular disorders) | 2 | 0
Venous thromboembolic event (Grade > =4) (Vascular disorders) | 2 | 1
Infusional reaction (General disorders) | 1 | 0
Infusion reaction Grade II (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Weakness (General disorders) | 1 | 0
Osteonecrosis of the jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain-musculoskeletal-joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Nail toxicity (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bilateral hand neuropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral neuropathy (Grade >=3) (Nervous system disorders) | 14 | 3
Peripheral neuropathy (Nervous system disorders) | 1 | 1
Peripheral neuropathy (motor or sensory) (grade >= 3) (Nervous system disorders) | 8 | 1
Sensory neuropathy (Nervous system disorders) | 1 | 0
Sensory neuropathy grade 2 (Nervous system disorders) | 1 | 0
Tingling in fingers grade I (Nervous system disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 2 | 0
Neuropathy of toes and clinical progression (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dizzy spells (Nervous system disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Epigastric pain (Gastrointestinal disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Recurrent right pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.